CLINICAL TRIAL: NCT00057317
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Dose-ranging Study to Determine the Efficacy, Safety, Tolerability and Pharmacokinetics of Ro 205-2349 in Patients With Type 2 Diabetes Mellitus
Brief Title: Study of Ro 205-2349 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: WM16177
Record Dates: First submitted 2003-03-31; First posted 2003-04-01 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: Ro 205-2349

SUMMARY:
The objective of the study is to determine the dose(s) of Ro 205-2349 which, when compared to placebo, are efficacious, safe and tolerable in improving glycemic control in patients with type 2 diabetes. Doses of 5 to 20 mg/day will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 75
* Type 2 diabetes for longer than 3 months
* HbA1c (glycosylated hemoglobin A1c) greater than 7.0% at screening
* FPG (fasting plasma glucose) greater than 126 mg/dL at screening
* BMI (body mass index) less than 40 kg/square meter

Exclusion Criteria:

* Type I diabetes
* Type 2 diabetes patients currently treated with insulin
* Type 2 diabetes patients currently or previously treated with Actos, Avandia or Rezulin
* FPG (fasting plasma glucose) greater than 270 mg/dL at baseline
* Impaired liver or kidney function
* Triglycerides greater than 600 mg/dL
* Uncontrolled hypertension
* Pregnant or lactating women
* Women not using adequate contraception

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (101):
- United States (60):
  - Huntsville, Alabama
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Encino, California
  - Fountain Valley, California
  - Fremont, California
  - Fresno, California
  - Irvine, California
  - Modesto, California
  - Pasadena, California
  - San Bruno, California
  - Santa Rosa, California
  - Sunnyvale, California
  - Hamden, Connecticut
  - Norwalk, Connecticut
  - Newark, Delaware
  - Hollywood, Florida
  - Jacksonville, Florida
  - Ocala, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Lawrenceville, Georgia
  - Honolulu, Hawaii
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Trenton, New Jersey
  - Albuquerque, New Mexico
  - Buffalo, New York
  - New Hyde Park, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Morrisville, North Carolina
  - Portland, Oregon
  - Tualatin, Oregon
  - Camp Hill, Pennsylvania
  - Connellsville, Pennsylvania
  - Philadelphia, Pennsylvania
  - East Providence, Rhode Island
  - Greer, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Lebanon, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Edmonds, Washington
  - Wenatchee, Washington
- Bulgaria (3):
  - Pleven
  - Plovdiv
  - Sofia
- Canada (11):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Courtice, Ontario
  - Ottawa, Ontario
  - Windsor, Ontario
  - Laval, Quebec
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec
  - St. John's
- Estonia (3):
  - Tallinn
  - Tartu
  - Võru
- Latvia (4):
  - Ogre
  - Talsi
  - Tukums
  - Valmiera
- Lithuania (2):
  - Kaunas
  - Vilnius
- Mexico (6):
  - Guadalajara
  - Mexico City
  - Mérida
  - Monterrey
  - Pachuca, Hidalgo
  - Tijuana
- Panama City, Panama
- Ponce, Puerto Rico
- Romania (7):
  - Arad
  - Brasov
  - Bucharest
  - Galati
  - Ploieşti
  - Târgovişte
  - Târgu Mureş
- United Kingdom (3):
  - Bracknell
  - Nottingham
  - Plymouth